CLINICAL TRIAL: NCT03924427
Title: An Open-Label, Single-arm, Multi-Center, Phase 3 Study to Evaluate the Efficacy and Safety of BMS-986165 in Japanese Subjects With Moderate-to-Severe Psoriasis
Brief Title: An Investigational Study to Evaluate Experimental Medication BMS-986165 in Japanese Participants With Moderate-to-Severe Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM011-066
Record Dates: First submitted 2019-04-16; First posted 2019-04-23 (Actual); Results first posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — deucravacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BMS-986165 (Experimental): Given daily
  Interventions: Drug: BMS-986165

INTERVENTIONS:
Drug: BMS-986165 — Oral tablet administration

SUMMARY:
The purpose of this study is to investigate BMS-986165 given to Japanese participants with moderate-to-severe psoriasis.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

a. For participants with plaque psoriasis: i. Stable plaque psoriasis for at least 6 months ii. Moderate to severe disease iii. Candidate for phototherapy or systemic therapy b. Additional protocol-specified inclusion criteria apply for subjects with psoriatic arthritis, erythrodermic psoriasis, or generalized pustular psoriasis

Exclusion Criteria:

1. Guttate, inverse, or drug-induced psoriasis at Screening or Baseline
2. History of recent infection
3. Prior exposure to BMS-986165

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- Japan (27):
  - Local Institution - 0014, Nagoya, Aichi-ken
  - Local Institution, Toon-Shi, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - University of Occupational and Environmental Health, Japan, Kitakyushu, Fukuoka
  - Sapporo Skin Clinic, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Local Institution, Morioka, Iwate
  - Tokai University Hospital, Isehara, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - Kochi Medical School Hospital, Nakoku, Kochi
  - University Hospital - Kyoto Preferctural University of Medicine, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Mie University Hospital, Tsu, Mie-ken
  - Local Institution - 0004, Matsumoto, Nagano
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Nihon University Itabashi Hospital, Itabashi-ku, Tokyo
  - The Jikei University Hospital, Minato-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa, Tokyo
  - Japan Community Health Care Organization Tokyo Yamate Medical Center, Shinjuku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Teikyo University Hospital, tabashi City, Tokyo
  - Kumamoto University Hospital, Kumamoto
  - Local Institution - 0003, Osaka
  - Local Institution - 0012, Osaka

REFERENCES:
- [Derived] Okubo Y, Morita A, Imafuku S, Tada Y, Tsuritani K, Shao Y, Popmihajlov Z, Napoli A, Hippeli L, Habiro K, Ohtsuki M. Deucravacitinib, an Oral, Selective, Allosteric Tyrosine Kinase 2 Inhibitor, in Japanese Patients With Plaque Psoriasis: In-Depth Analysis of Efficacy and Safety in the Phase 3 POETYK PSO-4 Trial. J Dermatol. 2025 Jun;52(6):953-966. doi: 10.1111/1346-8138.17744. Epub 2025 Apr 30. PMID 40304108
- [Derived] Morita A, Imafuku S, Tada Y, Okubo Y, Habiro K, Tsuritani K, Banerjee S, Hoyt K, Kisa RM, Ohtsuki M. Deucravacitinib in plaque psoriasis: Safety and efficacy through 3 years in Japanese patients in the phase 3 POETYK PSO-1, PSO-4, and LTE trials. J Dermatol. 2025 May;52(5):761-772. doi: 10.1111/1346-8138.17685. Epub 2025 Mar 11. PMID 40066907
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Deucravacitinib 6 mg QD: Deucravacitinib (BMS-986165) 6 mg once daily (QD)
Period: Overall Study
Arm/Group | Deucravacitinib 6 mg QD
Started | 74
Completed | 68
Not Completed | 6
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Deucravacitinib 6 mg QD
Number analyzed (Participants) | 74
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (11.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 57
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese | 73
  Asian - Non-Japanese | 1

OUTCOME MEASURES:

1. Primary Outcome: Static Physician's Global Assessment (sPGA) 0/1 Response as a Number of Participants With a sPGA Score of 0 or 1 at Week 16
Description: The sPGA is a 5-point scale of an average assessment of all psoriatic lesions based on erythema, scale, and induration. sPGA 0/1 is the response as a number of participants who experience a sPGA score that determines psoriasis severity as clear (0) or almost clear (1) with at least 2-point improvement from baseline at week 16 using the non-responder imputation (NRI) method. The higher sPGA score denotes to more severe disease activity:
  * Clear (0)
  * Almost clear (1)
  * Mild (2)
  * Moderate (3)
  * Severe (4)
Time Frame: Week 16
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- Plaque Psoriasis 6 mg QD: Subgroup of the all treated population with plaque psoriasis that received Deucravacitinib (BMS-986165) 6 mg once daily (QD)
- Generalized Pustular Psoriasis 6 mg QD: Subgroup of the all treated population with generalized pustular psoriasis that received Deucravacitinib (BMS-986165) 6 mg once daily (QD)
- Erythrodemic Psoriasis 6 mg QD: Subgroup of the all treated population with Erythrodemic psoriasis that received Deucravacitinib (BMS-986165) 6 mg once daily (QD)
Arm/Group | Plaque Psoriasis 6 mg QD | Generalized Pustular Psoriasis 6 mg QD | Erythrodemic Psoriasis 6 mg QD
Number analyzed (Participants) | 63 | 3 | 8
Participants | 52 | 0 | 4

2. Primary Outcome: Psoriasis Area and Severity Index (PASI) 75 Response Assessed as a Number of Participants Who Achieve a 75% Improvement From Baseline in the PASI Score at Week 16
Description: PASI is a measure of the average redness, thickness, and scaliness of psoriatic skin lesions (each graded on a 0 to 4 scale; 0 = none to 4 = very severe), weighted by the area of involvement (head, upper extremities, trunk, and lower extremities). The PASI produces a numeric score that can range from 0 to 72, with higher PASI scores denoting more severe disease activity. PASI 75 is the response as a number of participants who experience at least a 75% improvement in PASI score as compared with the baseline value using the non-responder imputation (NRI) method.
Time Frame: Week 16
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Plaque Psoriasis 6 mg QD | Generalized Pustular Psoriasis 6 mg QD | Erythrodemic Psoriasis 6 mg QD
Number analyzed (Participants) | 63 | 3 | 8
Participants | 48 | 2 | 3

ADVERSE EVENTS:
Time Frame: Serious Adverse Events and Adverse Events were monitored from first dose to 30 days post last dose (Up to approximately 3 months). Participants were assessed for All Cause Mortality from their date of randomization until study completion (Up to approximately 23 months)
Arm/Group | Deucravacitinib 6 mg QD
All-Cause Mortality (participants affected / at risk) | 0/74
Serious Adverse Events (participants affected / at risk) | 5/74
Other Adverse Events (participants affected / at risk) | 40/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deucravacitinib 6 mg QD (N=74)
COVID-19 (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Normal pressure hydrocephalus (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Deucravacitinib 6 mg QD (N=74)
Constipation (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Nasopharyngitis (Infections and infestations) | 23
Periodontitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
Acne (Skin and subcutaneous tissue disorders) | 7
Psoriasis (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03924427/Prot_SAP_000.pdf